CLINICAL TRIAL: NCT00508157
Title: A 16-Week, Multicenter, Randomized, Open-label Study to Assess the Effects of Aripiprazole Versus Other Atypical Antipsychotics in the Treatment of Schizophrenic Patients With Metabolic Syndrome
Brief Title: A Phase 4 Study to Assess the Effects of Aripiprazole Versus Other Atypical Antipsychotics in the Treatment of Schizophrenic Patients With Metabolic Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN138-489; Eudract Number: 2007 001217 42
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Results first posted 2010-07-20 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Metabolic Syndrome; Schizophrenia
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia | interventions — Aripiprazole; Risperidone; Quetiapine Fumarate; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Aripiprazole
- B (Active Comparator)
  Interventions: Drug: Continued Antipsychotic (Risperidone or Quetiapine or Olanzapine)

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 5 to 30 mg, once daily, 16 weeks
  Other Names: Abilify; BMS-337039
  Arms: A
Drug: Continued Antipsychotic (Risperidone or Quetiapine or Olanzapine) — Tablets, Oral, According to summary of product characteristics (SmPC)
  Arms: B

SUMMARY:
258 patients who have been treated for at least 3 months with oral olanzapine, risperidone or quetiapine in the treatment of schizophrenia and currently presenting with metabolic syndrome, will be randomized to: i) aripiprazole for 16 weeks, with flexible dosing within a range of 10 to 30 mg once daily (QD); or ii) continue for 16 weeks on the same atypical antipsychotic treatment prior to the study enrollment.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* with schizophrenia being treated with olanzapine, risperidone, or quetiapine for at least 3 months
* with diagnosis of metabolic syndrome
* not treated for 1 of the parameters of metabolic syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- Local Institution, Brussels, Belgium
- Czechia (6):
  - Local Institution, Brno
  - Local Institution, Havířov
  - Local Institution, Hradec Králové
  - Local Institution, Prague
  - Local Institution, Přerov
  - Local Institution, Roudnice nad Labem
- France (7):
  - Local Institution, Fains-Véel
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (2):
  - Local Institution, Ellwangen
  - Local Institution, Werneck
- Greece (2):
  - Local Institution, Chania-Crete
  - Local Institution, Corfu
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Gyula
- Spain (2):
  - Local Institution, Oviedo, Principality of Asturias
  - Local Institution, Barcelona
- Local Institution, Wetzikon, Switzerland
- Local Institution, Izmir, Turkey (Türkiye)

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 125 participants were enrolled in this study; 73 were considered baseline failures and were not randomized.
Groups:
- Control Group: Olanzapine 5 mg and 10 mg, risperidone 1 mg and 4 mg, and quetiapine 100 mg and 200 mg oral tablets. Participants entered the study at the same dose as prior to randomization. Dose adjustments during the study were allowed within the dose range specified in the respective Summaries of Product Characteristics (SmPCs), according the investigator's judgment. Participants were treated for 16 weeks.
- Aripiprazole: Aripiprazole 5 mg, 10 mg, and 15 mg tablets: 5 mg once daily (QD) orally during the first week; 10 mg QD orally during the second week. Dosing was adjusted in 5 mg increments every 7 days within a range of 10 to 30 mg daily. Participants were treated for 16 weeks.
Period: Overall Study
Arm/Group | Control Group | Aripiprazole
Started | 26 | 26
Randomized Sample | 26 | 26
Safety Sample | 26 | 25 (1 participant was withdrawn from study prior to receiving study drug & excluded from safety sample.)
Completed | 24 | 23
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Subject Withdrew Consent | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject no longer met study criteria | 0 | 1
Not completed — Other known cause | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Aripiprazole | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10.47) | 43.9 (11.16) | 42.3 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 13 | 15 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 23 | 26 | 49
  Black/African American | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
Body Mass Index (BMI) category [Number; unit: Participants]
  < 30 kg/m2 | 7 | 13 | 20
  >=30 kg/m2 | 19 | 13 | 32
Waist Circumference Category [Number; unit: participants]
  ≤ 102 cm for Men/ ≤ 88 cm for Women | 1 | 2 | 3
  > 102 cm for Men/ > 88 cm for Women | 25 | 24 | 49
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m2] | 31.45 [19.0 to 42.8] | 31.31 [25.1 to 49.1] | 31.38 [19.0 to 49.1]
Fasting Non-High Density Lipoprotein (HDL) Cholesterol [Mean (Full Range); unit: mg/dL] — Non-HDL cholesterol was calculated as fasting Total Cholesterol minus fasting HDL Cholesterol.
  mg/dL | 173.1 [118 to 267] | 169.0 [110 to 268] | 171.0 [110 to 268]
Waist Circumference [Mean (Full Range); unit: cm] | 107.1 [90 to 136] | 107.1 [91 to 134] | 107.1 [90 to 136]
Weight [Mean (Standard Deviation); unit: kg] | 89.1 (15.06) | 91.6 (18.83) | 90.3 (16.93)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Fasting Non-high Density Lipoprotein (HDL) Cholesterol at Week 16
Description: Non-HDL cholesterol was calculated as fasting Total Cholesterol minus fasting HDL Cholesterol.
Time Frame: Baseline, Week 16
Population: Last Observation Carried Forward (LOCF) data set, Non-HDL measurements obtained after start of a treatment with a lipid-lowering agent were excluded; last measurement prior was used for LOCF analyses. Baseline data was carried forward for LOCF analysis for subjects for whom no on-treatment measurements for fasting non-HDL cholesterol was available.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 26 | 25
percent change | 10.06 (4.35) | -2.3 (3.85)
Statistical Analysis 1: Comparison: Control Group vs Aripiprazole; Null hypothesis: no difference in mean percent change from baseline in fasting non-HDLC between aripiprazole and the control group at Week 16; Test type: Superiority or Other; ANCOVA; ANCOVA model: log of on-treatment to baseline ratio = log of baseline value, treatment, previous antipsychotic; Mean Difference (Final Values) = -11.28, 95% CI 2-sided [-19.14 to -2.66] — Relative difference of Aripiprazole vs. Control Group in terms of (mean % change from baseline/100)+1

2. Secondary Outcome: Number of Participants Remaining on Metabolic Syndrome at Week 16
Description: Metabolic syndrome is defined as the presence of at least 3 out of the following Adult Treatment Panel III-A (ATP III-A) criteria (all of which are to be assessed at the same visit): waist >102 cm in males, >88 cm in females; blood pressure (BP) systolic BP ≥130 or diastolic BP ≥85 mm Hg; fasting HDL <40 mg/dL in males, <50 mg/dL in females; fasting triglycerides ≥150 mg/dL; fasting glucose ≥100 mg/dL, and/or the start of a treatment for any of the parameters of metabolic syndrome during the course of the study.
Time Frame: Week 16
Population: LOCF, Safety Sample For handling missing values, the metabolic syndrome is assumed to be ongoing unless there is enough data to support the resolution of the metabolic syndrome.
Measure: Number; unit: participants
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 26 | 25
participants | 22 | 16
Statistical Analysis 1: Comparison: Control Group vs Aripiprazole; null hypothesis: no difference between Aripiprazole and Control Group; Test type: Superiority or Other; Cochran-Mantel-Haenszel; A relative risk < 1 favors Aripiprazole over Control Group; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.54 to 1.06]

3. Secondary Outcome: Mean Percent Change From Baseline in Fasting Lipid Parameters Through Week 16
Description: Mean percent change from baseline in total cholesterol, low-density lipoprotein (LDL), HDL, and triglycerides.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: This measure was not analyzed because the study was terminated early and there were insufficient data to draw meaningful conclusions.
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change From Baseline for Fasting Glucose Levels Through Week 16
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: as for outcome 3
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Change From Baseline in Body Weight Through Week 16
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: as for outcome 3
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Median Change From Baseline in Body Mass Index (BMI) Through Week 16
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: as for outcome 3
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scale Through Week 16
Description: A CGI-S assessment (a 7-point scale to evaluate the severity of symptoms) was performed at baseline (1=normal; 7=among the most extremely ill patients). A decrease in value indicates improvement.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: as for outcome 3
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Change From Baseline in Subjective Well-Being Under Neuroleptics Scale (SWN-short Form) Through Week 16
Description: The SWN-short form is a 20-item self-report instrument that measures subjective well-being under neuroleptics. 10 positive and 10 negative items cover 5 health domains (subscales) (4 items each): emotional regulation, self-control, mental functioning, social integration, and physical functioning. Individual scores range from 1 (not at all) to 6 (very much). With negative item scores being reversed, Subscale scores range from 4 to 24 and Total score ranges from 20 to 120.
Time Frame: Baseline, Week 4, Week 8,Week 12, Week 16
Population: as for outcome 3
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mean Change From Baseline in the Impact of Weight on Quality of Life (IWQoL-Lite) Scale Through Week 16
Description: IWQoL-Lite is a 31-item self-report inventory to assess the impact of weight on quality of life among patients with obesity. Subscales include: Physical Function, Self Esteem, Sexual Life, Public Distress and Work. The rescaled IWQoL-Lite Total Score is determined by the sum of the 1 to 5 scores on all 31 items and rescaling this sum to a 0-100 scoring with 0=the poorest and 100=the best quality of life. A change of 7.8 to 12.0 points on the rescaled IWQoL-Lite Total Score=a meaningful improvement. A change of -4.5 to -7.6 on the rescaled IWQoL-Lite Total Score=a meaningful deterioration.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: as for outcome 3
Arm/Group | Control Group | Aripiprazole
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Control Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 9/25 | 2/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=25) | Control Group (N=26)
Blood cholesterol increased (Investigations) | 0 | 2
Anxiety (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Headache (Nervous system disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Following a review of all studies in development, a strategic decision was made to terminate this study due to slow accrual. Patients randomized and treated at the time of study termination could continue the study as per protocol until completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.